CLINICAL TRIAL: NCT00100087
Title: A Safety and Feasibility Study of the TheraSight(TM) Ocular Brachytherapy System for Treatment of Age-Related Macular Degeneration
Brief Title: Safety Study for Treatment of Wet Macular Degeneration Using the TheraSight(TM) Ocular Brachytherapy System
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Theragenics Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPD-07-01
Record Dates: First submitted 2004-12-22; First posted 2004-12-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-01

CONDITIONS: Macular Degeneration; Choroidal Neovascularization
Keywords: macular degeneration; brachytherapy; choroidal neovascularization; retinal degeneration; retinal diseases
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization; Retinal Degeneration; Retinal Diseases

INTERVENTIONS:
Device: Ocular Brachytherapy

SUMMARY:
The study will investigate the safety and feasibility of using the TheraSight(TM) Brachytherapy System for treatment of wet age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This is a multi-center randomized study of three doses of radiation (assigned 1:1:1) delivered by the TheraSight(TM) Brachytherapy System in participants with choroidal neovascularization (CNV) secondary to wet (exudative) AMD. Each participant receives a single dose of radiation delivered by one-time only brachytherapy. Participants are followed for three years after the radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older.
* Active primary or recurrent subfoveal CNV secondary to AMD with minimally classic or occult lesion, where an active lesion is defined as one or more of the following:

  a) An increase > 10% in lesion size (greatest linear dimension) on screening fluorescein angiography compared to previous fluorescein angiography no more than 180 days preceding screening visit
  * b) Subretinal hemorrhage associated with CNV within 90 days of screening visit.
  * c) Visual acuity loss > 1 Snellen line in screening visual acuity compared to previous visual acuity no more than 180 days preceding screening
* Lesion < 6 mm greatest linear dimension (GLD)
* Submacular blood must comprise less than 75% of the total lesion
* Subretinal fibrosis must comprise less than 25% of the total lesion
* Study eye best-corrected vision of 20/100 or poorer measured on an ETDRS chart (< 48 letters correct)
* Fellow eye best-corrected vision that is at least one line better on an ETDRS chart than the best-corrected vision of the study eye
* HbA1c < 6%
* Read and signed informed consent

Exclusion Criteria:

* Prior AMD therapy treatment, including but not limited to laser and photodynamic therapy.
* Current or planned participation in the next 180 days in other experimental trials involving treatment of neovascular AMD in the study eye, ocular devices, or trials involving treatment for ocular conditions other than AMD.
* Prior ophthalmic surgery for the study eye other than cataract extraction and/or capsulotomy. A minimum interval of 180 days must elapse between cataract extraction or capsulotomy and study enrollment.
* Likely need for cataract surgery in study eye during the 180 days following TheraSight(TM) System treatment.
* Presence of other eye diseases that could compromise visual acuity in the study eye or that, in the clinical judgment of the evaluating study ophthalmologist, might create special risk for the study participant.
* CNV due to other causes such as ocular histoplasmosis or pathologic myopia.
* Endstage fibrotic disciform lesions.
* Diabetes requiring diet modification, or medication, or insulin.
* Current history of malignancy (except participants having basal cell carcinoma that was treated successfully, or other malignancy operated on or treated and in remission for five years prior to inclusion in the trial).
* Hypertensive retinopathy.
* Major cardiovascular or cerebrovascular event within the last year; examples include congestive heart failure, myocardial infarction, and stroke.
* Inability to complete follow-up.
* Allergy to fluorescein dye.
* Previous radiation to the study eye.
* Pregnancy at time of surgical procedure.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-10

PRIMARY OUTCOMES:
Incidence of serious adverse events 30 to 270 days after treatment

SECONDARY OUTCOMES:
Serious adverse events occurring 9 months to 3 years after treatment
Reported adverse events occurring at any time after treatment
Feasibility of device use based on physician interviews and ultrasonography
Observation of retinal and angiographic appearance of CNV lesion and best-corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Theragenics Clinical Site, Atlanta, Georgia
  - Theragenics Clinical Site, Augusta, Georgia
  - Theragenics Clinical Site, Indianapolis, Indiana
  - Theragenics Clinical Site, Boston, Massachusetts
  - Theragenics Clinical Site, Newark, New Jersey
  - Theragenics Clinical Site, Raleigh / Durham, North Carolina